CLINICAL TRIAL: NCT06402409
Title: Workpackage 1: Baseline Prevalence and Implications of Multimorbidity for the Management of Spinal Pain Workpackage 2: The Influence of Multimorbidity Treatment Burden on Long-term Prognosis of Individuals With Spinal Pain
Brief Title: Exploring Multimorbidity in Patients With Spinal Pain
Status: Recruiting | Type: Observational
Sponsor: Jacob Christiansen Gandløse (Other)
Responsible Party: Sponsor-Investigator, Jacob Christiansen Gandløse, Principal investigator, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: F2023-169
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Back Pain; Neck Pain; Comorbidities and Coexisting Conditions
Keywords: Multimorbidity; Comorbidities; Comorbidity; Neck Pain; Back Pain; Spinal pain
MeSH Terms: conditions — Back Pain; Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: No treatment burden: Individuals scoring a total of 0 points on the Multimorbidity Treatment Burden Questionnaire, reflecting no perceived treatment burden.
- Group 2: Low treatment burden: Individuals scoring a total of below 10 points (but over 0) on the Multimorbidity Treatment Burden Questionnaire, reflecting low perceived treatment burden.
- Group 3: Medium treatment burden: Individuals scoring a total of between 10 and 22 points on the Multimorbidity Treatment Burden Questionnaire, reflecting medium perceived treatment burden.
- Group 4: High treatment burden: Individuals scoring a total of over 22 points on the Multimorbidity Treatment Burden Questionnaire, reflecting high perceived treatment burden.

SUMMARY:
Spinal pain is frequently accompanied by other chronic conditions (multimorbidity) and the predicted rise in multimorbidity prevalence emphasizes the need for studies to understand its impact on patients with chronic pain conditions.

Therefore the aims of the two studies are to:

Work package 1 - Determine prevalence of multimorbidity among patients with spinal pain referred to hospital outpatient clinics. Examine associations with relevant health-related factors and cover the significance of multimorbidity in the diagnostic process, referral patterns and healthcare utilization.

Work package 2: Examine the association between treatment burden arising from multimorbidity and patient prognosis in structured rehabilitation.

Across both work packages data will be derived from individuals initially referred to the Department of Rheumatology at Aalborg University Hospital (AaUH) or the Medical Spine Clinic in Silkeborg (MSCS).

DETAILED DESCRIPTION:
Background:

Spinal pain is frequently accompanied by other chronic conditions (multimorbidity) and the predicted rise in multimorbidity prevalence emphasizes the need for studies to understand its impact on patients with chronic pain conditions.

Objectives:

Work package 1: Determine prevalence of multimorbidity among patients with spinal pain referred to hospital outpatient clinics. Examine associations with various health-related factors and cover the significance of multimorbidity in the diagnostic process, referral patterns and healthcare utilization.

Work package 2: Examine the association between treatment burden arising from multimorbidity and patient prognosis in structured rehabilitation.

Methods:

The project consists of two work packages: A cross sectional study (Work package 1) and a prospective observational cohort study (Work package 2).

Across both work packages data will be derived from individuals initially referred to the Department of Rheumatology at Aalborg University Hospital (AaUH) or the Medical Spine Clinic in Silkeborg (MSCS). In work package 1 patients with scheduled appointments at the Departments are identified via the hospital's electronic booking system. Secure questionnaires are sent via E-Boks.

Data for the work packages will be collected through the hospital's electronic journal systems, patient-reported outcome measures (PROMs) and external danish registers. PROMS will be collected with REDCap at baseline and 3, 6, and 12 months after the initial consultation in the outpatient clinics. The patients' unique civil registration number (CPR) will be linked to external Danish registries facilitated by the Danish Civil Registration System (CRS).

Variables:

Electronic questionnaires: Name, CPR number, Marital status, Height and weight, Smoking and alcohol habits, and PROMS (elaborated elsewhere)

Medical records: Past and current medication use, referral source (general practitioner, specialist, hospital), Past treatment attempts (physiotherapy, chiropractic, etc.), Information on any scans performed (if any), Signs of radiculopathy, Number of consultations.

External registries:

* "The Danish Civil Registration System": Age, sex, Migration status, Vital status.
* "The Danish National Patient Registry": Concurrent diseases (ICD-10 codes), Period from referral date to treatment start date, Start and end dates of outpatient treatment.
* "The Danish National Prescription Registry": All dispensed medications from Danish pharmacies (ATC codes).
* "The Population Education Register": Highest completed level of education (short, medium, long)
* "DREAM database": Income status and public financial support.

Statistical considerations:

Work package 1: A cross-sectional study

Prevalence of multimorbidity and frequency of other diseases will be reported as percentages and total counts and presented in a table. Regression analysis will be emplyed to determine whether the number of chronic conditions or specific clusters of chronic conditions are associated with the primary outcome, EQ-5D-5L, other patient-reported measures, and use of healthcare services. Additionally, patients will be divided into groups categorized by the Multimorbidity Treatment Burden Questionnaire following the classification established by Duncan et al. These categories will divide participants into four distinct categories: no burden (score 0), low burden (score <10), medium burden (score 10-22), and high burden (score ≥22). Analysis of Covariance (ANCOVA) will be employed to determine whether there are statistically significant differences in EQ-5D-5L scores between the groups while accounting for potential confounding covariates. Individual plots will be generated to visually depict the distribution of patient scores on EQ-5D-5L and Brief Pain Inventory across the four groups.

Work package 2: An observational prospective cohort study

As in work package 1, patients will be categorized into groups based on their baseline treatment burden. Mixed model with repeated measures will be utilized to determine whether there are statistically significant differences in EQ-5D-5L scores and BPI-scores between groups over time (baseline, 3-6-12 months follow-up), while accounting for potential confounding covariates. Line graphs with error bars will be generated to visually depict the changes in EQ-5D-5L and BPI across the four groups.

For both workpackages missing data will be addressed by multiple imputation or other means if not deemed appropiate. The imputation model will be informed by existing literature and by a dropout analysis. In addition, the selection of covariates for inclusion in the statistical models will be guided by current evidence and clinical reasoning to account for potential confounding factors.

In assessing the prevalence of multimorbidity, it is defined as the presence of two concurrent chronic diseases in a single individual. To discern which ICD-10 codes correspond to chronic health conditions, a unique script has been devised. This script draws from previous studies, particularly those focused on determining multimorbidity prevalence, and incorporates recommendations from international consensus on multimorbidity measurement in research. The validation of ICD-10 codes in the Danish National Patient Registry (DNPR) and the Primary Care Referral Registry (PCRR) has been systematically conducted across various diagnoses and studies, affirming their accuracy for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or above
* Are diagnosed with neck or back pain
* Diagnosis is established by or confirmed by a rheumatologist (clinical expert opinion)
* Speak, read and understand Danish

Exclusion Criteria:

* Withdraw consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred with spinal pain to Aalborg University Hospital's Department of Rheumatology or the Medical Spine Clinic in Silkeborg during the recruitment time.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life | EQ-5D-5L will be collected at baseline, 3, 6, and 12 months of follow-up.
  The EQ-5D-5L questionnaire is a standardized measure of health-related quality of life recommended for multimorbidity research. The EQ-5D-5L assesses health status across five dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a five-point ordinal scale ranging from 1 (indicating no problems) to 5 (indicating extreme difficulties) The EQ-5D index score can be regarded as a continuous outcome and ranges from -0.624 to 1, with higher scores indicating better general health and quality of life.

SECONDARY OUTCOMES:
Brief Pain Inventory | BPI will be collected at baseline, 3, 6, and 12 months of follow-up.
  The Brief Pain Inventory (BPI) is considered the secondary outcome variable. The questionnaire assesses pain in two dimensions: pain intensity and pain interference with function, mood, sleep, and social life, and is a recommended core outcome measure in clinical trials of chronic pain. All items are scored from 0-10, with 0 indicating no pain or interference and 10 indicating worst imaginable pain/completely interference. Hence the sum 0-40 is averaged between the four items about pain intensity, and the sum 0-70 is averaged between the seven items about pain interference.

OTHER OUTCOMES:
Multimorbidity Treatment Burden Questionnaire (MTBQ) | MTBQ will be collected at baseline, 3, 6, and 12 months of follow-up.
  MTBQ is considered the exposure variable. It is a 10-item self-reported measure designed to assess the burden experienced by individuals with multiple health conditions. The ten items cover various aspects of treatment burden, such as managing own health, including self-monitoring and lifestyle changes, dealing with medication-related challenges (e.g., adherence and obtaining prescriptions), coordinating healthcare appointments, and managing dependency on others. Each item is scored on a scale ranging from 0 to 100. A higher total score on the questionnaire indicates a higher burden.
Selected items from work ability index | The selected items from WAI will be collected at baseline, 3, 6, and 12 months of follow-up.
  In this project, five items from the Work Ability Index will be considered as covariates. These include items 1, 2, 4, 5, and 6. Item 1 asks patients to rate their current work ability compared to their lifetime best (Likert scale ranging from 0-10). Item 2 asks patients to rate their work ability in relation to the physical and mental demands of the job (Likert scale ranging from very poor to very good). Item 4 asks patients to estimate their work impairment due to their health (ranging from "in my opinion, I am entirely unable to work" to "There is no hindrance/ I have no diseases"). Item 5 asks patients to indicate the number of sick days in the past 12 months (Ranging from "None at all" to "100-365 days"), while item 6 asks patients to give their own assessment of their work ability in 2 years (Ranging from "Unlikely" to "Certain").
Insomnia Severity Index | ISI will be collected at baseline, 3, 6, and 12 months of follow-up.
  To assess the patient's sleep quality, the Insomnia Severity Index (ISI) will be utilized. ISI includes seven questions that measure the severity of insomnia experienced over the past two weeks. Respondents assess the severity of difficulties in falling asleep, staying asleep, waking up too early, satisfaction with current sleep, as well as the degree of concern or anxiety caused by sleep problems. Additionally, the impact of sleep difficulties on daytime functioning and whether others notice any impairment related to the sleep issue are also addressed. A 5-point Likert scale (0-4) is used to rate the severity of each area based on the individual's experience. The total score ranges from 0 to 28, where a higher score indicates a greater severity of insomnia. ISI is considered a covariate.
EQ-5D-5L-VAS | EQ-5D-5L-VAS will be collected at baseline, 3, 6, and 12 months of follow-up.
  EQ-5D-5L-VAS is a 100mm visual analogue scale (VAS) used to assess self-rated health. On this scale, 0 represents the worst imaginable health, while 100 represents the best imaginable health. EQ-5D-5L-VAS is considered a covariate.
Patient Health Questionnaire | PHQ will be collected at baseline, 3, 6, and 12 months of follow-up.
  Symptoms of depression will be assessed using Patient Health Questionnaire 2 (PHQ-2), which includes the first two items of the PHQ-9. Patients responded to questions regarding their level of interest or pleasure in activities and feelings of depression or hopelessness over the past two weeks. Responses were scored from 0 to 3, resulting in a total score ranging from 0 to 6, with higher scores indicating higher symptoms of depression. PHQ-2 is considered a covariate.ating higher symptoms of depression. (46). PHQ-2 is considered a covariate.
Generalized Anxiety Disorder | GAD will be collected at baseline, 3, 6, and 12 months of follow-up.
  Symptoms of anxiety were assessed using the Generalized Anxiety Disorder 2 (GAD-2), which comprises the first two questions of the GAD-7. Patients rated their levels of nervousness, anxiety, or worry, along with their ability to control worrying over the past two weeks. Responses were scored from 0 to 3, resulting in a total score ranging from 0 to 6, with higher scores indicating more pronounced symptoms of anxiety. GAD-2 is considered a covariate.
Global rating of change | GROC will be collected at 3, 6, and 12 months of follow-up.
  The Global Rating of Change (GROC) is a patient-reported outcome measure (PROM) that asks patients to rate: 'How do you perceive your back/neck pain now, compared to before you began treatment?' They can respond on a 7-point Likert scale ranging from -3 (Much worse) to +3 (Much better). GROC is considered a covariate.

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

REFERENCES:
- [Background] Ahlstrom L, Grimby-Ekman A, Hagberg M, Dellve L. The work ability index and single-item question: associations with sick leave, symptoms, and health--a prospective study of women on long-term sick leave. Scand J Work Environ Health. 2010 Sep;36(5):404-12. doi: 10.5271/sjweh.2917. Epub 2010 Apr 7. PMID 20372766
- [Background] Rashid M, Heiden M, Nilsson A, Kristofferzon ML. Do work ability and life satisfaction matter for return to work? Predictive ability of the work ability index and life satisfaction questionnaire among women with long-term musculoskeletal pain. BMC Public Health. 2021 Mar 24;21(1):584. doi: 10.1186/s12889-021-10510-8. PMID 33761910
- [Background] Pedersen MH, Duncan P, Lasgaard M, Friis K, Salisbury C, Breinholt Larsen F. Danish validation of the Multimorbidity Treatment Burden Questionnaire (MTBQ) and findings from a population health survey: a mixed-methods study. BMJ Open. 2022 Jan 3;12(1):e055276. doi: 10.1136/bmjopen-2021-055276. PMID 34980626
- [Background] Duncan P, Murphy M, Man MS, Chaplin K, Gaunt D, Salisbury C. Development and validation of the Multimorbidity Treatment Burden Questionnaire (MTBQ). BMJ Open. 2018 Apr 12;8(4):e019413. doi: 10.1136/bmjopen-2017-019413. PMID 29654011
- [Background] Janssen MF, Pickard AS, Golicki D, Gudex C, Niewada M, Scalone L, Swinburn P, Busschbach J. Measurement properties of the EQ-5D-5L compared to the EQ-5D-3L across eight patient groups: a multi-country study. Qual Life Res. 2013 Sep;22(7):1717-27. doi: 10.1007/s11136-012-0322-4. Epub 2012 Nov 25. PMID 23184421
- [Background] Sorensen J, Davidsen M, Gudex C, Pedersen KM, Bronnum-Hansen H. Danish EQ-5D population norms. Scand J Public Health. 2009 Jul;37(5):467-74. doi: 10.1177/1403494809105286. Epub 2009 Jun 17. PMID 19535407
- [Background] Soer R, Reneman MF, Speijer BL, Coppes MH, Vroomen PC. Clinimetric properties of the EuroQol-5D in patients with chronic low back pain. Spine J. 2012 Nov;12(11):1035-9. doi: 10.1016/j.spinee.2012.10.030. PMID 23199409
- [Background] Walters SJ, Brazier JE. Comparison of the minimally important difference for two health state utility measures: EQ-5D and SF-6D. Qual Life Res. 2005 Aug;14(6):1523-32. doi: 10.1007/s11136-004-7713-0. PMID 16110932
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Song CY, Lin SF, Huang CY, Wu HC, Chen CH, Hsieh CL. Validation of the Brief Pain Inventory in Patients With Low Back Pain. Spine (Phila Pa 1976). 2016 Aug 1;41(15):E937-E942. doi: 10.1097/BRS.0000000000001478. PMID 26839985
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] Sapra A, Bhandari P, Sharma S, Chanpura T, Lopp L. Using Generalized Anxiety Disorder-2 (GAD-2) and GAD-7 in a Primary Care Setting. Cureus. 2020 May 21;12(5):e8224. doi: 10.7759/cureus.8224. PMID 32582485
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246